CLINICAL TRIAL: NCT03754686
Title: Oseltamivir Versus Paracetamol for Influenza-like Illness During the Influenza Season: a Randomized Controlled Trial
Brief Title: Oseltamivir Versus Paracetamol for Influenza-like Illness During the Influenza Season
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0520-18-RMB CTIL
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oseltamivir (Active Comparator): best medical care and oral oseltamivir 75 mg twice daily for five days.
  Interventions: Drug: Oseltamivir
- Paracetamol (Active Comparator): best medical care and oral paracetamol twice daily for five days.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Oseltamivir — Best medical care and oral oseltamivir 75 mg twice daily for five days. Dose adjustments of oseltamivir will be made according to manufacturer's instructions.
  Arms: Oseltamivir
Drug: Paracetamol — Best medical care and oral paracetamol twice daily for five days
  Other Names: Best medical care and oral paracetamol twice daily for five days.
  Arms: Paracetamol

SUMMARY:
Parallel group, investigator initiated, 1:1, open-label, non-inferiority randomized controlled trial, aiming to show that paracetamol is non-inferior to oseltamivir among patients with serious acute respiratory infection (SARI).

DETAILED DESCRIPTION:
Study setting: a single tertiary hospital, containing 1,000 beds. Intervention: best medical care and oral oseltamivir 75 mg twice daily for five days.

Control: best medical care and oral paracetamol twice daily for five days. Dose adjustments of oseltamivir will be made according to manufacturer's instructions. Patients with creatinine clearance between 30-60 ml/minute will receive 30 mg twice daily for five days. Patients with creatinine clearance 10-30 ml/minute will receive 30 mg, once daily for 5 days. Hemodialytic patients will receive 30 mg upon admission, and 30 mg after every session, for 5 days. Patients on peritoneal dialysis will receive 30 mg once, which suffices for 5 days. Patients may withdraw participation from the trial at any time. The attending physician may also be informed the treatment arm, and start antiviral treatment if deemed necessary.

A nasopharyngeal swab for influenza will be obtained upon enrollment. PCR testing will be performed in-house. Administration of oseltamivir or paracetamol for patients with negative swabs will be stopped, unless the sample was obtained after initiation of the study drug. Patients may discontinue or refuse trial medications at any point. The reasons for discontinuation will be documented.

Adverse effects: The investigators will monitor and document daily rate of nausea, vomiting, and headache, deterioration in kidney function (defined as an increase in creatinine by >0.3 mg/dl or by >50% from baseline), and in-hospital delirium.

Participant timeline and follow-up: After signing informed consent (available in Hebrew, Arabic or Russian), study personnel, will interview patients and review electronic medical files.

Patients enrolled will be followed-up daily by study personnel in-hospital, until the first of: achieving clinical improvement (defined below), hospital discharge, or 7 days from randomization. During the follow-up patients will be assessed for clinical improvement and for AE (detailed above). Patients discharged before day 7 will be assumed to have reached clinical improvement by that time. Readmissions and deaths by day 30 will be monitored through the electronic patient file (Prometheus), providing access to a national registry of hospitalizations and updated from the national Health Ministry on deaths.

Recruitment: during the influenza high-season, ER nurses will fill in a check-box containing the SARI criteria items. An electronic report of all cases filling SARI criteria, will be sent to study personnel 5 times daily. An investigator will apply inclusion and exclusion criteria on candidates, and obtain informed consent from patients or their legal guardians. Enrollment will continue until reaching the predefined sample size.

Randomization and blinding methods: a computer-generated randomizer will be used, to assign all patients into block sizes of 8, with a 1:1 randomization rate. Allocation codes will be concealed in sealed opaque envelopes that will be opened consecutively by the randomization code. The study is open-label. Outcome assessment will be performed blinded to the treatment allocation.

Patients will be assessed once daily, by study personnel, for the clinical course of the disease and for AE. Data will be entered into a case report form (CRF). Daily assessment will end when patients are released from hospitalization, or at the end of 7 days from admission. During hospitalization, medical files will be reviewed for administration of antibiotics, respiratory deterioration (defined as new requirement of oxygen supplementation or requirement for mechanical ventilation, either invasive or non-invasive). Duration of hospitalization, as well as re-hospitalization within one month after enrollment, and 30 days mortality, available from the hospital computerized medical records, will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* admitted to the hospital during the influenza "high season" with SARI.

Exclusion Criteria:

1. Severe disease on admission, defined as any of the following: patients deemed to require intensive care immediately upon admission, a high probability of imminent respiratory failure as judged by the ER physician.
2. Pregnancy.
3. Severe immunosuppression including: Acquired immunodeficiency syndrome (AIDS) or Human immunodeficiency virus (HIV) with unknown CD4 or with CD4 < 200/mL, solid organ and stem cell transplant recipients, or neutrophil count of less than 100 per µliter.
4. Patients with decompensated cirrhosis.
5. Patients discharged home from the ER.
6. Patients unable to sign informed consent with no legal guardian.
7. Patients who received at least 2 doses of oseltamivir prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2019-02-10 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
the composite of failure to reach clinical stability at day 7 after randomization OR transfer to the ICU until day 7 after randomization OR re-admission within 30 days of randomization OR death within 30 days of randomization. | 30 days
  Clinical stability will be defined as: heart rate < 100/min AND systolic blood pressure > 90 mmHG AND temperature ≤ 38.00 AND respiratory rate ≤ 24 AND oxygen saturation ≥ 90.

SECONDARY OUTCOMES:
include time to clinical stability (defined earlier), and duration of hospitalization. | 30 days

IPD SHARING:
Plan to Share IPD: No